CLINICAL TRIAL: NCT05035082
Title: REALYSE - Comparative Effectiveness of Once-daily Oral Semaglutide Versus Any Other Oral Glucose-lowering Medication in a Real-world Adult Population With Type 2 Diabetes on Metformin Monotherapy in US Based Health Care Systems - a Pragmatic Randomized Trial
Brief Title: A Research Study Comparing RYBELSUS® to Other Blood Sugar Lowering Tablets in People Living in America With Type 2 Diabetes (REALYSE)
Acronym: REALYSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4558; U1111-1253-2577 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- oral semaglutide (Experimental): All participants are given tablets used in addition to metformin.
  Interventions: Drug: semaglutide
- other oral glucose lowering medication (Active Comparator): All participants are given tablets used in addition to metformin.
  Interventions: Drug: oral glucose-lowering medications (commercially available)

INTERVENTIONS:
Drug: semaglutide — Oral administration The doctor will give a prescription for the medicine and tell how to take it.
  Arms: oral semaglutide
Drug: oral glucose-lowering medications (commercially available) — Oral administration The doctor will give a prescription for the medicine and tell how to take it.
  Arms: other oral glucose lowering medication

SUMMARY:
This study is comparing the medicine RYBELSUS® to other medicines in people with type 2 diabetes who need extra treatment. All medicines used in this study are tablets which lower blood sugar in people with type 2 diabetes. The purpose of the study is to see how well RYBELSUS® is at lowering blood sugar compared to other tablets when used in addition to metformin. Participants doctor will give participants either RYBELSUS® or any other blood sugar lowering tablets - which treatment participants get is decided by chance. The doctor treating participants diabetes will give participants a prescription for the medicine and tell how to take it. The study will last for about 1 year. Participants will have 2 planned visits with their doctor which are part of the usual routine diabetes management: the first visit is when participants are included in the study, the second visit is a 1-year follow-up visit. In addition, the study personnel will contact participants up to 3 times during this period and to follow-up on information from participant doctors visits. Participant will be asked to respond 3 times to 4 questionnaires via their personal smartphone or tablet or paper if participant do not have access to one during the study. All clinic visits are part of the usual routine diabetes management and are covered by participants health insurance plan. The study team will collect information from these visits recorded in the medical chart. Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Key inclusion criteria

* Treatment with metformin as monotherapy prior to eligibility assessment that has failed to result in adequate glycemic control at the discretion of the investigator or treatment provider. However, prior short-term treatment with an oral glucose lowering agent or insulin for up to 14 consecutive days in addition to metformin is allowed if discontinued prior to screening.
* Current member of a health plan which includes pharmacy benefits.
* HbA1c greater than or equal to 7% within last 90 days prior to the day of screening or to be taken before randomization.
* Further intensification with an additional glucose-lowering oral agent including oral semaglutide is indicated according to approved prescribing information to achieve glycemic target at the discretion of the treatment provider.

Key exclusion criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using contraception.
* Any disorder which in the investigator's or treatment provider's opinion might jeopardize patient's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated hemoglobin A1c (HbA1c) | From randomization to year 1
  percentage-points

SECONDARY OUTCOMES:
Patient achieving HbA1c below 7.0% (Yes /No) | Year 1
  Count of patient(s)
Patient achieving HbA1c below or equal to 6.5% (Yes/No) | Year 1
  Count of patient(s)
Patient achieving HbA1c below 7.0% or at least 1.0%-point reduction in HbA1c (Yes/No) | From randomization to year 1
  Count of patient(s)
Patient achieving greater than or equal to 5% reduction in body weight (Yes/No) | From randomization to year 1
  Count of patient(s)
Patient achieving individualized HbA1c target per Healthcare Effectiveness Data and Information Set (HEDIS) criteria (below 8.0% if age greater than or equal to 65 years or with defined comorbidities or otherwise below 7.0%) (Yes/No) | Year 1
  Count of patient(s)
Patient achieving HbA1c less than or equal to treatment provider defined individualized target (Yes/No) | Year 1
  Count of patient(s)
Relative change in body weight (%) | From randomization to year 1
  Percentage
Change in body weight (lbs) | From randomization to year 1
  Lbs
Time to treatment intensification (add-on) or change (switch) | From randomization to year 1
  Days
Diabetes Treatment Satisfaction Questionnaire, change version (DTSQc), Relative treatment satisfaction total score | Year 1
  Score on a scale (The Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) will be used to measure the change in patient satisfaction with their diabetes treatment. It consists of a six-item scale assessing treatment satisfaction and two items assessing perceived frequency of hyperglycaemia and hypoglycaemia. The DTSQc items are on a scale from 3 to -3. If they experience no change, then 0 is chosen. Higher score indicate higher satisfaction with their current treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (25):
- United States (25):
  - Stewart Medical Group, Alhambra, California
  - FDRC, Costa Mesa, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Raincross Medical Group, Riverside, California
  - Reyes Clinical Research, Inc, Miami, Florida
  - DC Research Works, Marietta, Georgia
  - Urban Family Practice Assoc, Marietta, Georgia
  - Macoupin Research Group, Gillespie, Illinois
  - UnityPoint Health-Diabetes Care Center, Peoria, Illinois
  - Endeavor Health, Skokie, Illinois
  - Kernodle Clin Dpt-Pvt Diagnost, Burlington, North Carolina
  - OnSite Clinical Solutions, LLC_Charlotte, Charlotte, North Carolina
  - WakeMed Garner Hlthplx, Garner, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Central Ohio Clinical Research LLC, Columbus, Ohio
  - Jefferson Endocrinology Assocs, Philadelphia, Pennsylvania
  - Tristar Clin Investigations, PC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians_Pittsburgh, Pittsburgh, Pennsylvania
  - AnMed Health IMA, Anderson, South Carolina
  - Baylor Scott & White Res Inst, Dallas, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - DCT-Stone Oak, San Antonio, Texas
  - Chrysalis Clinical Research, St. George, Utah

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com